CLINICAL TRIAL: NCT05527197
Title: What do Patients Report Regarding Their Real-world Function Following Combined First MTP and First TMT Arthrodesis?
Brief Title: Patient Reported Function Following Combined First MTP and First TMT Arthrodesis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Bunion Center, LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Double Joint Arthrodesis
Record Dates: First submitted 2022-05-11; First posted 2022-09-02 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-09

CONDITIONS: Hallux Valgus
Keywords: Bunion
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patient reported function of daily ADL's post combined first MTP/TMT joint arthrodesis (Other): Patients that meet the inclusion criteria will be contacted for participation in the study. If the patient agrees to participate in the study, informed consent will be obtained. The retrospective study will consist of a chart review and baseline radiographic analysis. The prospective follow-up will consist of the patient completing the Post-Operative Function and Satisfaction Survey via phone call with study staff. Radiographic images will be analyzed by a single central radiologist.
  Interventions: Device: Lapiplasty

INTERVENTIONS:
Device: Lapiplasty — The Lapiplasty® System instruments and implants will be retrospectively evaluated in patients previously surgically treated with the Lapiplasty® Procedure for Triplane MTP and TMT joint arthrodesis.
  Other Names: Treace Medical Concepts, Inc

SUMMARY:
The goal of the study is to gather sufficient patient data to assess real world postoperative function after a first metatarsophalangeal (MTP) joint arthrodesis done in conjunction with first tarsometatarsal arthrodesis (TMT) (double fusion). Many studies have demonstrated the success of a first MTP joint arthrodesis in eliminating pain and reducing the intermetatarsal angle. Very little research has been published to assess the outcomes of double arthrodesis. Limited research has specifically assessed patients' everyday function and gait following MTP arthrodesis and no studies are available to assess real world function following double arthrodesis. More data that includes patient reported function during activities of daily living is needed to understand the benefits and draw backs of combined first MTP/TMT joint arthrodesis used to treat and correct first ray deformity.

DETAILED DESCRIPTION:
* Retrospective clinical data will be collected on a Clinical Data Collection Form from a chart abstraction at the research site.
* All radiographs will be anonymized and transferred in a secure process to a Central Radiologist for the study. The data will be collected in excel spreadsheet or on a Radiographic Data Collection Form.
* Post-operative function and satisfaction will be collected by study personnel via telephone call with the patient
* De-identified data will be entered into a database for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with surgeon identified indications for double joint arthrodesis
2. Previous double joint arthrodesis procedure (Lapiplasty® Procedure) between 2017-2021
3. Procedure completed at least 12 months from the onset of the study
4. Early weight-bearing protocol (< 3 weeks)
5. Patients between 18 and 80 years of age, inclusive at the time of the procedure
6. Clinical and radiographic follow up available at least 6 months post double joint arthrodesis procedure
7. Willing to answer the Post-Operative Functional and Satisfaction Questionnaire via phone call

Exclusion Criteria:

1. Diabetes with neuropathy
2. Presence of previous infection of operative foot
3. Documented neuropathy of any cause
4. Concomitant hindfoot or ankle procedures except tendon procedures or Gastrocnemius recession

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Patient reported level of activity and satisfaction based on functional surveys | 12 months post procedure
  Patient responses in the Double Arthrodesis Sports Activities Related to Operative Foot Questionnaire and Sports Activities Related to Operative Foot Questionnaire

SECONDARY OUTCOMES:
Comparison of Pre-Operative and Post-Operative Radiographic Alignment | Baseline, 6 months post procedure
  X-ray comparison of operative foot
Radiographic Assessment of Healing of first Metatarsophalangeal (MTP) Joint Arthrodesis | 6 months post procedure
  1. Appropriate radio density and trabecular pattern at joint arthrodesis interface
  2. No lucency at joint arthrodesis
Clinical Assessment of Healing of first Metatarsophalangeal (MTP) Joint Arthrodesis | 6 months post procedure
  1. Absence of clinical motion
  2. Absence of pain at the arthrodesis site
Clinical Assessment of Healing of first Tarsometatarsal (TMT) Joint Arthrodesis | 6 months post procedure
  1. Absence of clinical motion
  2. Absence of pain at the arthrodesis site
Radiographic Assessment of Healing of first Tarsometatarsal (TMT) Joint Arthrodesis | 6 months post procedure
  1. Appropriate radio density and trabecular pattern at joint arthrodesis interface
  2. No lucency at joint arthrodesis
Time to start of weight-bearing in boot | 0-3 weeks
  The time needed for a study subject to begin bearing weight in a boot after the procedure
Time to start of weight-bearing in shoe | 0-12 weeks
  The time needed for a study subject to begin bearing weight in a shoe after the procedure
Time to return to full unrestricted activity, | 6 weeks to 12 months
  The time needed for a study subject to return to full unrestricted activity after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Dayton DPM FACFAS, Principal Investigator — Foot & Ankle Center of Iowa
Locations (1):
- Foot and Ankle Center of Iowa, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No